CLINICAL TRIAL: NCT03938675
Title: Early Use of Mother's Own Raw Milk, Maternal Satisfaction, and Breastfeeding Continuation in Hospitalised Neonates: A Prospective Cohort Study
Brief Title: Early Use of Raw Milk and Breastfeeding Continuation
Acronym: DOAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: DOAL
Record Dates: First submitted 2019-04-09; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Breastfeeding Continuation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Raw maternal own milk before day 7: Without any intervention, investigators observed whether neonates received raw MOM during the first week of life. Accordingly, the neonates were grouped as "exposed" when they received any raw MOM before day 7, versus "unexposed" when they did not receive any raw MOM before day 7.
- No Raw maternal own milk before day 7: Without any intervention, investigators observed whether neonates received raw MOM during the first week of life. Accordingly, the neonates were grouped as "exposed" when they received any raw MOM before day 7, versus "unexposed" when they did not receive any raw MOM before day 7.

SUMMARY:
BACKGROUND:

Despite the critical importance of breast milk for preterm and sick neonates, there is no consensus regarding the use of raw mother's own milk (MOM) in neonatal units.

OBJECTIVES:

This study aimed to describe the use of raw MOM in hospitalised neonates before day 7 (early use), and to investigate: (i) related factors, (ii) maternal satisfaction, and (iii) the association with breastfeeding continuation.

METHODS:

This prospective cohort included 516 neonates intended to be breastfed in 2 French neonatal units. Neonates receiving raw MOM before day 7 were compared to those who did not. The association between early use of MOM and breastfeeding continuation at hospital discharge, and up to 6 months later, was measured by logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Eligible neonates were those admitted between April 2012 and June 2013, who were intended to be breastfed and remained hospitalized for 7 days or more.

Exclusion Criteria:

* Neonates with parents not fluent in French were excluded.

Max Age: 6 Months | Sex: All
Age Groups: Child
Study Population: Neonates male or female admitted between April 2012 andJune 2013, who were intended to be breastfed and remained hospitalized for 7 days or more.
Sampling Method: Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Change in breastfeeding after hospital discharge | On Day 60 and Day 180 after hospital discharge
  Breastfeeding was defined as the consumption of any mother's own milk (MOM), provided either directly at the breast or after having been expressed. Information on breastfeeding continuation was extracted from the electronic chart during the last 2 days preceding hospital discharge. It was classed as "exclusive" when all the fed milk was MOM, or "partial" when it was completed by other milk and/or food.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Laborie, MD, Principal Investigator — Hospices Civils de Lyon